CLINICAL TRIAL: NCT03196700
Title: Short Course Accelerated Radiation Therapy in Palliative Treatment of Advanced Head and Neck Malignancies
Brief Title: Short Course Radiation Therapy in Palliative Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHARON-H&N
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Palliative Care
Keywords: palliative care; head and neck cancer; radiotherapy; pain; quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Short course radiotherapy (Experimental): The radiotherapy is delivered over two days with accelerated hypo-fractionation was delivered
  Interventions: Radiation: Short course radiotherapy

INTERVENTIONS:
Radiation: Short course radiotherapy — An accelerated hypo-fractionation radiotherapy is delivered for palliation in patients with metastatic or locally advanced head and neck cancer.

SUMMARY:
The study wants to define the maximum tolerated dose (MTD), safety and efficacy of a short course radiation treatment in patients with symptomatic advanced head and neck cancer.

DETAILED DESCRIPTION:
The study wants to define the maximum tolerated dose (MTD) of a conformal short course accelerated radiation therapy delivered in twice daily fractions and 2 consecutive days, and the feasibility of this fractionation in term of safety and efficacy for symptomatic palliation of metastatic or locally advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven locally advanced or metastatic H&N cancer
* excluded from curative therapy because of disease stage and/or presence of multiple comorbidities and/or poor performance status
* age > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status < 3

Exclusion Criteria:

* prior RT to the same region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 1 year
  The maximum tolerated dose is defined as the dose level below the highest administered dose associated with dose limiting toxicity (DLT) in at least one third of patients

SECONDARY OUTCOMES:
Acute toxicity | 1 year
  Acute toxicity after treatment is evaluated with CTCAE scale
Quality of life | 1 year
  Quality of life after the treatment is evaluated according to CLAS scale
Pain relief | 1 year
  Pain after the therapy is evaluated with the visual analogic scale
Late toxicity | 1 year
  Late toxicity after the treatment is evaluated with EORTC-RTOG scale

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G. Morganti, MD, Principal Investigator — Radiation Oncology Center, Department of Experimental, Diagnostic and Specialty Medicine - DIMES, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided